CLINICAL TRIAL: NCT05944029
Title: Therapeutic Effects of Pomegranate Seed Powder on Metabolic Syndrome Markers
Brief Title: Effect of Pomegranate Seed Powder on Markers of Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asif Ali (Other)
Responsible Party: Sponsor-Investigator, Asif Ali, Researcher, University of Veterinary and Animal Sciences, Lahore - Pakistan
Organization: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UVAS
Record Dates: First submitted 2023-04-11; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Hypertension; Obesity; Insulin Resistance; Diabetes; Pomegranate seed powder; Dyslipidemia
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Obesity; Insulin Resistance; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Prospective Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic syndrome Patients (Experimental): Pomegranate seed powder is administered for alleviating symptoms of metabolic syndrome
  Interventions: Dietary Supplement: Pomegranate seed powder

INTERVENTIONS:
Dietary Supplement: Pomegranate seed powder — 10 g powder / day
  Other Names: Punica granatum

SUMMARY:
Metabolic syndrome is a public health concern worldwide and in Pakistan as well. Abdominal obesity, hyperglycemia, hypertriglyceridemia, hypertension, and low HDL cholesterol are its hallmarks while pomegranate seed's unique chemical composition has sparked research into the health benefits in same arena as weight control, blood lipid profile changes, and other metabolic disturbances. It's high time to study therapeutic efficiency of Pomegranate seed powder against metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic syndrome, accumulation of certain metabolic risk factors, such as abdominal obesity, hyperglycemia, hypertriglyceridemia, hypertension, and low HDL cholesterol, has been noted as one of the most important risk factors for the epidemic of type 2 diabetes and cardiovascular disease in the 21st century. It has become a significant public health concern and a global epidemic with a prevalence rate of about 25% among American adults. Multiple researches have demonstrated the effectiveness of pomegranate in the management of diabetes, inflammatory conditions, obesity, and blood lipid levels, and consequently metabolic syndrome. Various pomegranate components have the potential to substitute anti-diabetic medications as well Pomegranate seed's unique chemical composition has sparked research into the health benefits, such as weight control, blood lipid profile changes, and other metabolic disorders.

seed powder can influence the patient's metabolic syndrome-related indicators.

Hypothesis:

Pomegranate seed powder can be effective to treat the individuals with impaired metabolism.

Methodology:

In a clinical trial, patients of metabolic syndrome (n=50) will be given pomegranate seed powder dose for over 8 weeks, twice a day. Biochemical outcomes including blood pressure, FBG, cholesterol, hemoglobin level will be determined before and after the completion of trial in addition to patient's weight. Finally, using one-way ANOVA and T-test, collected data will be analyzed.

Expected outcome: The study will explore the potential of pomegranate seed powder in treating metabolic syndrome's risk factors. Therefore, our findings on the studied parameters of patient will assist future researchers in developing tested, evidence-based recommendations.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25kg/m2
* Dyslipidemia
* Altered blood glucose level
* Age 30-55 ( male and female)

Exclusion Criteria:

* Thyroid disorder
* Liver disease
* Kidney disorder
* Cancer etc

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-08-24 (Estimated)

PRIMARY OUTCOMES:
Lipid Profile | 7 weeks
  The change in Lipid Profile, after consuming Pomegranate seed powder for 7 weeks will be assessed, to look for improvements.
Fasting Glucose | 7 weeks
  The change in Blood Glucose level, after consuming Pomegranate seed powder for 7 weeks will be assessed, to look for improvements.
Blood Pressure | 7 weeks
  The change in both systolic and diastolic blood pressure after consuming Pomegranate seed powder for 7 weeks will be assessed, to look for improvements.
Weight | 7 weeks
  The change in weight, after consuming Pomegranate seed powder for 7 weeks will be assessed, to look for improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Asif Ali, Mphil, Study Director — University of Veterinary and Animal Sciences Lahore
Locations (1):
- University of Veterinary and Animal sciences Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Intervention study, data will be confidential to maintain patients privacy, enrollment of patients with their consent

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT05944029/Prot_SAP_ICF_000.pdf